CLINICAL TRIAL: NCT04026620
Title: The Trajectory of Fetal Alcohol Spectrum Disorders (FASD) Across the Life Span: Continuing Prevention and Longitudinal Epidemiology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: University of Stellenbosch (Other); University of New Mexico (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 12-1827; 5R01AA015134 (NIH)
Record Dates: First submitted 2019-07-17; First posted 2019-07-19 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-08

CONDITIONS: Fetal Alcohol Spectrum Disorders
Keywords: alcohol use and abuse; prenatal alcohol use
MeSH Terms: conditions — Fetal Alcohol Spectrum Disorders; Alcohol Drinking

STUDY DESIGN:
Intervention Model Description: A total of 400 women who screen positive for drinking will be asked if they want to be enrolled in the efficacy trial. Once a participant enrolls into the efficacy trial study, they are then randomly assigned to either the MET (Motivational Enhancement Therapy) group or informational pamphlet-only group. The MET group will be provided: 1.) a one (1) hour and 30 minute MET session, 2.) an information pamphlet on FASD written in simple Afrikaans. Women in the control condition will receive two informational pamphlets (one on FASD advising abstinence from alcohol use and one describing fetal development, both in Afrikaans). The data obtained by nurses during a woman's initial prenatal clinic visit for all 400 participants (Self-administered Questionnaire and AUDIT), will be matched with deliveries of the newborns to monitor the birth outcomes of newborns of participating mothers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pamphlet-only (Other): Pamphlet-only women will be provided with two (2) informational pamphlet(s) (both in Afrikaans).
  Interventions: Behavioral: Informational Pamphlet
- MET Group (Other): MET women will be provided with a one (1) hour and 30 minute session of Motivational Enhancement Therapy (MET) and informational pamphlet(s) (both in Afrikaans).
  Interventions: Behavioral: Informational Pamphlet; Behavioral: Brief Motivational Enhancement Therapy (MET) Session

INTERVENTIONS:
Behavioral: Informational Pamphlet — The control group will be provided with two (2) informational pamphlets (and have it read to those who are of lower literacy). Pamphlets contain information about the harmful effects of drinking alcohol during pregnancy and the harmful effects of alcohol on the unborn baby.
Behavioral: Brief Motivational Enhancement Therapy (MET) Session — The case control trial/efficacy study will provide a one-session MET session in Afrikaans (the predominant language of the region). The face-to-face session will provide information to help people and pregnant women who want to change their drinking behavior, become 'dry' and stay motivated to change their drinking behaviors. Sessions will be approximately one (1) hour and 30 minutes.
  Arms: MET Group

SUMMARY:
Screen women of childbearing age (15 - 44 years) for high risk drinking in antenatal clinics of the established research sites in the Western Cape Province of South Africa (SA). While there are multiple reasons for this screening, the purpose is for selective (secondary) prevention of FASD. A.) Initiate a case control trial/efficacy study (n=400) of the use of one-session brief motivation enhancement therapy (MET) in busy public health settings (versus information only) in these rich research sites where very high rates of FASD have been documented over the entirety of the past two decades. B.) These targeted prevention activities follow both findings and staff experience in prevention over the past decade which indicate that the most likely venue for prevention activities is in antenatal clinics of the local, primary care clinics and hospitals. These activities will also provide tangible community-level pay back for participation in ongoing research activities and lay the groundwork for sustainable services going forward.

DETAILED DESCRIPTION:
The purpose of the research is to find out if Motivational Enhancement Therapy is more effective than printed information alone (Informational pamphlets only) in helping women reduce their risk of giving birth to children with Fetal Alcohol Spectrum Disorders (FASD) at Primary Health Care Facilities, in addition to evaluation individuals for risky health behaviors by having them complete brief screening questionnaires that give them information of how much risk they might be facing from their alcohol or other drug use. When a pregnant mother drinks alcohol, she puts her baby at risk. FASD is a group of growth, mental, and physical problems that may occur in a baby when a mother drinks alcohol during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Drinking pregnant women who are defined as women who:

  * Drank in the 3 months prior to pregnancy and/or
  * Drank alcohol at least once at any time during the prenatal period.
* Gestational age less than or equal to 16 weeks, but not more than 20 weeks at intake

Exclusion Criteria:

* Non-drinking pregnant women who are defined as women who have not had any alcohol during the past 30 days.
* Gestational age >20 weeks

Ages: 15 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 167 (Actual)
Dates: Start 2019-08-06 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip A May, Ph.D., Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Stellenbosch University, Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pamphlet-only | MET Group
Started | 82 | 85
Completed | 71 | 68
Not Completed | 11 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pamphlet-only | MET Group | Total
Number analyzed (Participants) | 82 | 85 | 167
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.3 (6.2) | 26.5 (6.9) | 26.4 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 85 | 167
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 82 | 85 | 167
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 0 | 0 | 0
  More than one race | 80 | 83 | 163
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  South Africa | 82 | 85 | 167

OUTCOME MEASURES:

1. Primary Outcome: Change in the Alcohol Use Disorders Identification Test (AUDIT) Score Over Time
Description: The AUDIT is a 10-item, self-report, screening tool to assess alcohol consumption, drinking behaviors, and alcohol-related problems. The AUDIT was developed and adopted by the World Health Organization. AUDIT scoring for questions 1 to 8 are scored on a five-point scale from 0,1,2,3, or 4; questions 9 and 10 are scored on a three-point scale from 0,2, or 4. The minimum total score for the AUDIT is 0. The maximum total score for the AUDIT is 40. Interpretation of the AUDIT Total Score is as follows: 0-7 indicates a low-risk level; a score of 8-15 is risky or hazardous level; a score of 16-19 is a high-risk or harmful level; and 20 or more is considered high-risk/almost certainly dependent on alcohol.
Time Frame: Baseline through 9 months post-partum, an average of approximately 67 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pamphlet-only | MET Group
Number analyzed (Participants) | 71 | 68
score on a scale | -5.8 (6.7) | -4.0 (7.5)

ADVERSE EVENTS:
Time Frame: From the time of signing informed consent through nine months post-partum, on average, approximately 67 weeks total.
Arm/Group | Pamphlet-only | MET Group
All-Cause Mortality (participants affected / at risk) | 0/82 | 0/85
Serious Adverse Events (participants affected / at risk) | 0/82 | 0/85
Other Adverse Events (participants affected / at risk) | 0/82 | 0/85

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-26): https://cdn.clinicaltrials.gov/large-docs/20/NCT04026620/Prot_SAP_000.pdf